CLINICAL TRIAL: NCT02600598
Title: Biological Effects of LEO 43204 in Actinic Keratosis Assessed by Histopathology
Brief Title: Biological Effects of LEO 43204 in Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0084-1228
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2018-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 Group A (Experimental): Group A - Experimental LEO 43204, applied once daily for 3 consecutive days in patients with actinic keratosis
  Interventions: Drug: LEO 43204 Gel, 0.037%
- LEO 43204 Group B (Experimental): Group B - Experimental LEO 43204, applied once daily for 3 consecutive days in patients with actinic keratosis
  Interventions: Drug: LEO 43204 Gel, 0.037%

INTERVENTIONS:
Drug: LEO 43204 Gel, 0.037%
  Arms: LEO 43204 Group A
Drug: LEO 43204 Gel, 0.037%
  Arms: LEO 43204 Group B

SUMMARY:
This is a Phase I, single-centre, open label, within-subject comparison trial to explore the biological effects of LEO 43204 Gel, 0.037%, applied once daily for 3 consecutive days in patients with actinic keratosis on the upper extremity. The treatment area for each patient will be as defined as a contiguous area of 250 cm2 of skin on the upper extremity (including the dorsum manus) that contains a minimum of 5 AK lesions. Additionally there must be at least one AK lesion located in a non-treated area on the contralateral arm. All eligible subjects will receive LEO 43204 Gel, 0.037%, on the treatment area on Days 1, 2 and 3. Study medication application will be (sub)investigator applied. A total of 30 patients will be enrolled into this study (n=15 in each of the two groups). Patients will be divided into two groups with different biopsy schedules.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed and dated informed consent has been obtained.
* 2. Subjects with at least 5 non-keratotic, clinically typical, visible and discrete AK lesions within a contiguous 250 cm2 area (AK Treatment Area) on the upper extremity,
* 3. Subjects with one additional AK lesion located on the contralateral arm.
* 4. Subjects with an area of normal skin in close proximity to the AK Treatment Area or on the contralateral arm.
* 5. Male and female subjects, 18 years or older.
* 6. Agreement from the patient to allow photographs of the selected treatment area to be taken and used as part of the study data package
* 7. Ability to follow study instructions and likely to complete all study requirements
* 8. Female Subjects must be of either

  * non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus or has tubal litigation) or,
  * child-bearing potential* provided there is a confirmed negative pregnancy test prior to trial treatment to rule out pregnancy.

    * Female subjects are considered of child-bearing potential unless they have had a hysterectomy or have undergone tubal litigation or have been post-menopausal for at least one year prior to first visit.
* 9. Female subjects of child-bearing potential must be willing to use effective contraception at trial entry and until completion.

Effective contraception is defined as follows:

* Abstinence (when this is in line with the preferred and usual life style of the subject).
* Vasectomised partner (given that the subject is monogamous).
* An intrauterine device.
* Double barrier method defined as two distinct methods (two actual barrier methods).
* Hormonal contraceptive (oral hormonal birth control, oestrogenic vaginal ring, percutaneous contraceptive patches, implants and injectables) for at least one menstrual cycle prior to enrolment.

Exclusion Criteria:

* 1. Prior treatment with ingenol mebutate gel in the treatment area within the last 12 months.
* 2. Previously assigned treatment in this clinical trial or previously participated in a clinical trial in the LEO 43204 programme (presently LP0084-68, LP0084-1013, LP0084-1014, LP0084-1015, LP0084-1148, LP0084-1077, LP0084-1193, LP0084-1194, LP0084-1195, LP0084-1196).
* 3. Location of the selected treatment area within 5 cm of an incompletely healed wound or infected area of the skin (excl. study related biopsies) or within 5 cm of a suspected basal cell carcinoma (BCC) or SCC.
* 4. History or evidence of skin conditions other than the study indication that would interfere with the histologically- or biomarker evaluation of the study medication (e.g. eczema, unstable psoriasis, xeroderma pigmentosum).
* 5. Treatment area lesions that have an atypical clinical appearance (e.g. hypertrophic, hyperkeratotic, recalcitrant disease [had cryosurgery on two previous occasions] and/or cutaneous horns).
* 6. Known sensitivity or allergy to any of the ingredients of LEO 43204 Gel (e.g. citric acid)
* 7. Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety during the course of the study, as determined by Investigator clinical judgment.
* 8. Anticipated need for in-patient hospitalisation or in-patient surgery during the study period. Note that cosmetic/therapeutic procedures are not excluded if they fall outside of the criteria detailed in the Prohibited Therapies or Medications (listed below).
* 9. Anticipated excessive or prolonged exposure to ultraviolet light (e.g. sunlight) or use of tanning beds for the duration of the study
* 10. Current participation in any other interventional clinical trial
* 11. Subjects who have received treatment with any non-marketed drug product (i.e. an agent which has not yet been made available for clinical use following registration) within the last two months.
* 12. Subjects known to be infected with Human Immunodeficiency Virus (HIV).
* 13. Subject known or, in the opinion of the investigator, is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state).
* 14. Females who are pregnant, of child-bearing potential and wishing to become pregnant during the trial, or are breast feeding.
* 15. Females of child-bearing potential with positive pregnancy test at [screening or visit 1].
* 16. Previous enrolment in this clinical trial. Prohibited Therapies and/or Medications: within 2 weeks prior to the Screening visit
* 17. Cosmetic or therapeutic procedures (e.g. use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing): within 2 cm of the selected treatment areas and within 2 cm of the selected AK lesion outside the treatment area
* 18. Use of acid-containing therapeutic products (e.g. salicylic acid or fruit acids, such as alpha and beta hydroxy acids and glycolic acids), topical retinoids or light chemical peels: within 2 cm of the selected treatment areas and within 2 cm of the selected AK lesion outside the treatment area
* 19. Use of topical salves (non-medicated/non-irritant lotion/cream are acceptable) or topical steroids: within 2 cm of the selected treatment areas and within 2 cm of the selected AK lesion outside the treatment area; artificial tanners: within 5 cm of the selected treatment areas and within 5 cm of the selected AK lesion outside the treatment area Prohibited Therapies and/or Medications: within 4 weeks prior to the Screening visit
* 20. Treatment with immunomodulators (e.g. azathioprine), cytotoxic drugs (e.g. cyclophosphamide, vinblastine, chlorambucil, methotrexate, podophyllin, camptothecin) or interferon/interferon inducers.
* 21. Treatment with systemic medications that suppress the immune system (e.g. cyclosporine, prednisone, methotrexate, infliximab).
* 22. Treatment/therapy with UVB

Prohibited Therapies and/or Medications: within 8 weeks prior to the Screening visit

* 23. Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 2 cm of the selected treatment areas and within 2 cm of the selected AK lesion outside the treatment area Prohibited Therapies and/or Medications: within 6 months prior to the Screening visit
* 24. Use of systemic retinoids (e.g. isotretinoin, acitretin, bexarotene)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12-27 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Number of CD3+ T lymphocytes assessed by immunohistochemistry in biopsies from AK lesions 56 days after first treatment. | 56 days

SECONDARY OUTCOMES:
Number of infiltrating cells assessed by immunohistochemical staining | 8 weeks
Expression of inflammatory and skin matrix modulation markers assessed by RNA expression and immunohistochemistry | 8 weeks
Expression of ICAM-1 (marker of vascular endothelium activation) assessed by immunohistochemical staining as area of section with positive staining. | 8 weeks
Expression of Ki-67 and K16 (markers of cell proliferation and differentiation) assessed by immunohistochemical staining as area of section with positive staining. | 8 weeks
Expression of cleaved caspase-3 (apoptosis) assessed by immunohistochemical staining as area of section with positive staining | 8 weeks
Necrosis of the epidermis and dermis in haematoxylin & eosin-stained sections (scored on 0-3 scale). | 8 weeks
Number of p53 gene mutations determined by DNA sequencing in normal and AK skin and blood at baseline and in a treated AK lesion at Week 8. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Siegel, MD, Principal Investigator — Long Island Skin Cancer and Dermatology Surgery
Locations (2):
- United States (2):
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Long Island Skin Cancer and Dermatology Surgery, Smithtown, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en